CLINICAL TRIAL: NCT04460638
Title: SARS-CoV2 (COVID-19) Diagnosis in Human Saliva by MALDI-TOF MS Profiling
Acronym: CoviDiagMS
Status: Completed | Type: Observational
Sponsor: Direction Centrale du Service de Santé des Armées (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-COVID19-15; 2020-A01249-30 (Other: IDRCB)
Record Dates: First submitted 2020-07-06; First posted 2020-07-07 (Actual); Last update posted 2023-09-06 (Actual); Status verified 2023-09

CONDITIONS: SARS-CoV 2
Keywords: MALDI-TOF MS

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Saliva samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Covid+ hospitalization group: Patients hospitalized with SARS-CoV2 infection
  Interventions: Biological: Saliva collection; Other: Clinical assessment
- Covid+ outpatient group: Patients or caregivers followed on an outpatient basis for an SARS-CoV2 infection
  Interventions: Biological: Saliva collection; Other: Clinical assessment
- Covid- group: Caregivers not infected with an SARS-CoV2
  Interventions: Biological: Saliva collection; Other: Clinical assessment
- Non-SARS pathology group: Individuals not infected with SARS-CoV2 but with another acute and/or infectious non-SARS pathology
  Interventions: Biological: Saliva collection; Other: Clinical assessment

INTERVENTIONS:
Biological: Saliva collection — Saliva samples are regularly collected over a period of up to 30 consecutive days.
Other: Clinical assessment — The participant's clinical data will be collected regularly over a period of up to 30 consecutive days.

SUMMARY:
Since March 2020, SARS-CoV2 virus (nCoV19; COVID-19) is considered pandemic. Its high rate of spread and infection in the human population and the lack of effective and validated treatment have led the authorities of several countries to confine their populations to slow the spread of COVID-19. As part of the management of this health crisis, the screening of individuals is essential in order to isolate "infected cases". These screening tests are currently performed on nasopharyngeal swabs using RT-PCR for the detection of viral RNA. Although sensitive and specific, these tests remain relatively long (2-5 hours), expensive and the strong international demand for nucleic extraction kits and enzymes are factors limiting the implementation of widespread screening (problem of supply of swabs, molecular biology consumables).

In order to prevent the risks of a shortage of screening means, we propose to develop an innovative alternative strategy, PCR-free, based on the detection of specific protein signatures in human saliva by MALDI-TOF MS profiling. MALDI-TOF MS profiling is a method used in routine diagnostics by microbiology laboratories for the identification of microorganisms. MALDI-TOF MS profiling has been successfully used to classify individuals according to their infectious status (oral pathologies) based on the analysis of their saliva, but also as a tool for the identification of respiratory viruses from cell culture supernatants. In addition, we have expertise and skills in the field of MALDI-TOF MS profiling and have implemented new strategies to improve the quality of profiles and their analysis, particularly in the context of entomological and vector identification projects. Finally, recent Chinese studies have reported that COVID-19 was detectable in saliva by RT-PCR.

The main objective of this study is to develop a test based on the MALDI-TOF profiling method to detect individuals infected with SARS-CoV2 from saliva sample.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age;
* screened for SARS-CoV2 by RT-PCR from a nasopharyngeal swab within 96 hours prior to inclusion.

Exclusion Criteria:

* Patient admitted to intensive care;
* Pregnant woman.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population consists of patients and caregivers infected and uninfected with CoV2-SARS.
Sampling Method: Non-Probability Sample
Enrollment: 779 (Actual)
Dates: Start 2020-07-23 (Actual); Primary Completion 2021-08-13 (Actual); Study Completion 2021-08-13 (Actual)

PRIMARY OUTCOMES:
Development of a test based on the MALDI-TOF profiling method to detect individuals infected with SARS-CoV2 from saliva sample. | Day 30
  The development of this test is based on machine learning techniques, which involve "training" a mathematical model, in which the results of the mass spectrometry analysis of saliva samples and clinical data will be used to determine the information needed to distinguish a saliva sample from a SARS-CoV2-infected participant from a healthy saliva sample.

SECONDARY OUTCOMES:
Rate of correct classification by the test (MALDI-TOF MS profiling) from saliva sample | Day 30
  For each saliva sample, the status ("correct" or "incorrect") of the classification of the sample ("infected" or "not infected") by the test (MALDI-TOF MS profiling) will be determined. Then the rate of correct classification will be calculated. The test will be considered efficient when it has reached a correct classification rate of more than 95%.
Rate of correct classification by RT-PCR from saliva sample | Day 30
  For each saliva sample, the status ("correct" or "incorrect") of the classification of the sample ("infected" or "not infected") by RT-PCR will be determined. Then the rate of correct classification by RT-PCR will be calculated.
Identification of proteins specific to the SARS-CoV2 infection | Day 30
  On each saliva sample, the expression of proteins will be determined using mass spectrometry. By comparison between SARS-CoV2 infected saliva samples and non-infected saliva samples, the presence of proteins that are specifically expressed in SARS-CoV2 infected saliva samples will be determined.
Presence of a positive anti-SARS-CoV2 antibody response by RT-PCR | Day 30
  On each SARS-CoV2 infected saliva sample, the presence of anti-SARS-CoV2 antibodies, by RT-PCR, will be determined.
Correlation between the identified protein markers and the clinical course of the participants. | Day 30
  In SARS-CoV2 infected participants (Covid+ hospitalization group and Covid+ outpatient group), the presence of a correlation between the presence of proteins specific to the SARS-CoV2 infection and the clinical evolution of patients will be determined.

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital d'Instruction des Armées Laveran, Marseille, France

IPD SHARING:
Plan to Share IPD: Undecided